CLINICAL TRIAL: NCT01034722
Title: Fat Globules in Breast Milk
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Prof' Nachum Vaisman, Tel Aviv Sourasky Medical Center
Other Study IDs: TASMC-09-NV-593-CTIL
Record Dates: First submitted 2009-12-16; First posted 2009-12-17 (Estimated); Last update posted 2009-12-17 (Estimated); Status verified 2009-11

CONDITIONS: Fat Globules in Breast Milk
Keywords: Breast Milk; Fat Globules

STUDY DESIGN:
Observational Model: Ecologic or Community
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Western Diet: Volunteer mothers with western diet.
- Vegetarians: volunteer mothers with vegetarians diet
- Bedouins: Volunteer mothers who are Bedouins

SUMMARY:
The aims of this study is:

1. To investigate the diet influence on size and composition of fat globules in breast milk under controlled diet.
2. To study the changes in globules distribution along one session of lactation and during the day.

Study design:

Subjects:

This will be a open label study. Each subject will serve as his own control. Study population will include 45 volunteer mothers, that will divide to 3 groups: 15 vegetarians, 15 western diet and 15 Bedouins.

Each participant will be nursing a 2-5 months baby. Each participant will sign an informed consent. Each participant will be ask to collect 2 milk samples twice a day i.e.- once on the first nursing in the morning (in the beginning and at the end of the nursing session), and once in the evening on last nursing again, (in the beginning and at the end). Each sample will contain 5 ml of milk.

Participants will be asked to repeat the procedure one month later.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteers nursing only babies aged 2-5 months.
* Age: 20-45 years old.
* Written informed consent.

Exclusion Criteria:

* Nursing babies more than 5 months or less than 2 months.
* Infants who consume breast milk replacement formulas on top of breast milk.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Study population will include 45 volunteer mothers, that will divide to 3 groups: 15 vegetarians, 15 western diet and 15 Bedouins.
  Each participant will be nursing a 2-5 months baby.
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2009-12; Primary Completion 2010-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
To investigate the diet influence on size and composition of fat globules in breast milk under controlled diet.
To study the changes in globules distribution along one session of lactation and during the day.

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Medical Center, Tel Aviv, Israel